CLINICAL TRIAL: NCT04295629
Title: Research on the Effects of Ilioinguinal Nerve Block on Chronic Pain in Patients Who Undergo Inguinal Hernia With Spinal Anesthesia
Brief Title: The Effects of Ilioinguinal Nerve Block on Chronic Pain in Patients in Inguinal Hernia With Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tugba Onur, Principle İnvestigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-17/24
Record Dates: First submitted 2020-02-29; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Ilioinguinal Nerve Block
Keywords: Inguinal hernia; Ilioinguinal nerve block; Chronic Pain
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: 60 ASA I-III patients between ages 18-65 who underwent single-sided inguinal hernia operation were randomly classified into two groups in the operating room as; Group I (n:30); spinal block (SA), Group 2 (n:30); SA and ilioinguinal block (IHNB). All patients were given SA in sitting position and 3ml 0.5% hyperbaric bupivacaine was injected in sterile conditions with 25 G injection in L3-4, L4-5 subarachnoid space. Times when the block reached T10 level were recorded. Ultrasoundguided ilioinguinal block was implemented and 10 ml 5% bupivacaine was injected to patients in group I with peripheric nerve block injection in the reanimation unit after the surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VAS (Visüel Analog Score) (Active Comparator): VAS : 0-10 points 0 means: no pain 10 means: incredible pain
  Interventions: Procedure: Research on the effects of Ilioinguinal Nerve Block on Chronic Pain in Patients who undergo Inguinal Hernia with Spinal Anesthesia; Procedure: Ilioinguinal nerve block
- LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) (Active Comparator): LANSS 0-24 points >12 points : has chronic neuropathic pain <12 points: no chronic neuropathic pain
  Interventions: Procedure: Research on the effects of Ilioinguinal Nerve Block on Chronic Pain in Patients who undergo Inguinal Hernia with Spinal Anesthesia; Procedure: Ilioinguinal nerve block

INTERVENTIONS:
Procedure: Research on the effects of Ilioinguinal Nerve Block on Chronic Pain in Patients who undergo Inguinal Hernia with Spinal Anesthesia — The patients underwent inguinal hernia operation randomly classified into two groups in the operating room as; Group I (n:30); spinal block (SA): All patients were given SA in sitting position and 3ml 0.5% hyperbaric bupivacaine was injected in sterile conditions with 25 G injection in L3-4, L4-5 subarachnoid space. Times when the block reached T10 level were recorded.
  Other Names: Spinal Anesthesia
Procedure: Ilioinguinal nerve block — Group 2 (n:30); SA in sitting position and 3ml 0.5% hyperbaric bupivacaine was injected in sterile conditions with 25 G injection in L3-4, L4-5 subarachnoid space and as a ilioinguinal block (IHNB) 10 ml 5% bupivacaine was injected to patients with peripheric nerve block injection in the reanimation unit after the surgery.

SUMMARY:
Regional anesthesia is a popular anesthetic method in patients who will undergo an inguinal hernia operation. Researchers known that pain in the operating area is a complaint that impairs the quality of life for patients in the long term after the operation. In addition to regional anesthesia, has planned to investigate the effects of applying another drug near the surgery area on pain that may develop in the long term.

DETAILED DESCRIPTION:
Post-operative chronic pain can be defined as the neuropathic-characterized pain persisting at least 3 months after the surgery despite healing of the operation area.

However, it is still uncertain if the underlying physio-pathologic mechanism is due to intraoperative direct nerve injury or it is resulting from indirect nerve injury caused by inflammatory mesh. Post-operative chronic pain restricts the daily activities, causes anxiety and depression, increases use of analgesics and imposes a serious economic burden by increased use of health services and medical treatment. For this reason, today post-operative chronic pain is considered as an important complication of surgery. Researchers can list the risk factors of pain development as; age, weight, preoperative and postoperative pain, surgical method, recurrence, anesthesia method. Various oral non-steroid and/or opioid agents have been used in chronic pain treatment but nowadays interest in regional anesthesia approaches is increasing due to increased systemic side effects. Aim in this study is to evaluate the effects of postoperative ilioinguinal block implementation on chronic pain in patients who will undergo inguinal hernia operation with spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-65
* Inguinal hernia operation with spinal anesthesia
* Patients who agreed to participate in the study

Exclusion Criteria:

* Mental retards and communication disorder
* Infection at the injection site
* Patient with a clotting disorder
* Local anesthetic allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
acute pain scores( VAS) | 24 hours
  Presence of pain was interrogated in the hospital within the first 24 hours (2nd, 6th, 12th, 24th hours), Visüel Analog Scale (VAS) is between 0-10 points, 0 means no pain and 10 means incredible pain.
chronic pain scores(LANSS) | 6 months
  The presence of pain that may occur in the 3rd and 6th months can be learned by contacting patients by phone. The Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) is a neuropathic pain scale. In LANSS follow-ups, 12 points or more were associated with neuropathic pain.

SECONDARY OUTCOMES:
taken amount of analgesic drugs | 48 hours
  compared how many milligram analgesic agents are given to the patient will be followed.
postoperative complications | 48 hours
  compared complications such as nausea, vomiting, motor or sensorial disorder after 48 hours of operation
hospital stay | 48 hours
  compared how many days patients stayed in the hospital until they were discharged

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Onur, MD, Principal Investigator — 2017-17/24
Locations (1):
- University of Health Sciences Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No